CLINICAL TRIAL: NCT04617587
Title: Structural Variations of the Neural Genome as Prognostic Biomarkers for Prematurity Related Neurodevelopmental Disorders in Childhood
Brief Title: Novel Epigenetic Biomarker for Prematurity Related Neurodevelopmental Disorders in Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Ministero della Salute, Italy (Other); Istituto Nazionale di Genetica Molecolare, Milan Italy (Unknown); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR-2018-12365280
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Premature Birth
Keywords: Premature Birth; DNA Methylation; L1 Elements; Epigenometics; Early Intervention; Brain Development; Neurodevelopment; Parent-infant interaction; Massage therapy; Visual interaction
MeSH Terms: conditions — Premature Birth | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Intervention (Experimental): All the enrolled preterm infants are assigned to receive the early neurodevelopmental intervention during the NICU stay.
  Interventions: Behavioral: Early Intervention

INTERVENTIONS:
Behavioral: Early Intervention — The early intervention (EI) is delivered during the NICU stay. It is a multisensory intervention which consists in three parts: parental training, massage therapy and visual interaction. The EI is first focused on parental training, according to PremieStart Protocol, in order to train parents to: recognize signs of infant stress and alert-available behavior through the identification of infant's behavioral states; adopt principles of graded stimulation; sustain infant's attention and respond to infant's cues; optimize interactions and avoid overwhelming infants through facilitation strategies. The program is held in eight main sessions and one additional post-discharge session. In addition, parents are trained and invited to daily promote preterm baby massage therapy and visual interaction (visual fixation/tracking and visual attention).

SUMMARY:
Preterms are early exposed to a stressful environment (i.e. excessive sensory stimulation and paucity of parental contact) with subsequent detrimental effects on brain maturation and neurodevelopmental outcomes. In contrast, early interventions seem to reduce stress exposure and promote neurodevelopment. The brain functional plasticity in response to environmental experiences can be partly attributed to changes in DNA methylation. In this context, LINE-1 (L1) promoter (18% of human genome) methylation/demethylation has been associated with L1 somatic mobilization in the brain genomes, contributing to experience-driven brain plasticity; this mechanism being deregulated in important neurological disease. This study aims at identifying and characterizing the role of L1 DNA repeats as a novel biomarker to predict long-term neurodevelopmental outcome in preterm infants. In addition, the study's secondary goal will be to define a preventive approach, based on early intervention strategies, for improving long-term neurodevelopmental outcomes.

DETAILED DESCRIPTION:
Around 25-50% of very preterm infants suffer from neurodevelopmental delays (motor, cognitive and behavioral problems), which are most likely related to brain micro-structural defects and impaired neuronal maturation and connectivity. These alterations in brain maturation occurring during the neonatal period may be implicated in long-term neurobehavioral disorders later experienced by preterm babies.

There is increasing evidence that also stressful events (excessive sensory stimulation, paucity of parental contact and painful procedures) experienced in the Neonatal Intensive Care Unit (NICU) by preterm neonates can affect neurodevelopment through epigenetic mechanisms.

The brain is a genomic mosaic, owing to somatic mutations that arise throughout development. It is already established that mobile genetic elements, including LINE-1 (L1), are one source of somatic mosaicism, inducing copy number variations in neural genome. Environmental experiences can drive brain plasticity at a molecular level, with changes in DNA methylation. In particular, L1 promoter methylation/demethylation is already associated with L1 mobilization in the brain genomes and its deregulation is linked with important neurological diseases. A preliminary study has shown the correlation between L1 promoter methylation levels and preterm birth. In addition, maternal care during early life has been reported to drive variability in L1 mobilization and methylation of the neural hippocampal genome in mice models.

Several studies have reported how individualized developmental care in the NICU can ameliorate preterm infants' medical outcome and subsequent neurodevelopment. More recently, early intervention (EI) strategies based on parental training and multisensory stimulation, such as infant massage and visual stimulation, have been demonstrated to enhance child's neurodevelopment. These programs have the greatest potential to reduce environmental stress in preterms, promoting brain plasticity, optimizing dyadic interaction and ameliorating neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth between 24+0 and 32+6 weeks
* Mothers age over 18 years
* Good comprehension of the Italian language
* Written informed consent signed by both parents

Exclusion Criteria:

* Infants with major genetic disorders and malformations
* Parents declined study participation
* Single-parent family
* Parents with obvious cognitive or psychiatric disorders and drug addiction

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
L1 Promoter Methylation Levels on Biological Materials | Up to 24 months corrected age
  Epigenetic analysis is performed on biological materials: cord blood sample and buccal swab at birth, peripheral blood sample and buccal swab at NICU discharge/term equivalent age, buccal swab collected during the follow up assessment at 12 and 24 months of corrected age.

SECONDARY OUTCOMES:
Conventional and advanced brain Magnetic Resonance Imaging (MRI) | Term equivalent age, approximately 40 weeks postmenstrual age
  Evaluation of brain development and maturation
Neurological Examination | Term equivalent age, approximately 40 weeks postmenstrual age
  Hammersmith Neonatal Neurological Examination (HNNE)
General Movements Examination | Term equivalent age, approximately 40 weeks postmenstrual age
  Prechtl's Qualitative Assessment of General Movements
Visual Assessment | Term equivalent age, approximately 40 weeks postmenstrual age
  Neonatal Visual Assessment Battery developed by Ricci et al. The assessment evaluates the following items: ocular spontaneous motility, ability to fix and follow a target, reaction to colour, visual acuity and visual attention at distance.
Neurodevelopmental Outcome | Up to 24 months corrected age
  Children development assessed using the Griffiths Mental Development Scales, performed at 12 and 24 months of corrected age. Mean score is 100. General score has a Standard deviation of 12 and sub scales have a Standard Deviation of 16.
  Higher scores indicate better outcomes.
Behavioral Outcome | 24 months corrected age
  Children behavior assessed using the Child Behavior Checklist (CBCL). It is a parent report form to screen for emotional, behavioral and social problems.
  Lower scores indicate better outcomes. A T score above 75 is considered pathological while a T score between 65 and 74 is considered borderline.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Fumagalli, MD, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Beatrice Bodega, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- NICU, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The dataset generated for this study will be made available on request in an anonymized version or in a grouped form in order to prevent patient identification.

REFERENCES:
- [Background] Fontana C, De Carli A, Ricci D, Dessimone F, Passera S, Pesenti N, Bonzini M, Bassi L, Squarcina L, Cinnante C, Mosca F, Fumagalli M. Effects of Early Intervention on Visual Function in Preterm Infants: A Randomized Controlled Trial. Front Pediatr. 2020 Jun 4;8:291. doi: 10.3389/fped.2020.00291. eCollection 2020. PMID 32582595
- [Background] Newnham CA, Milgrom J, Skouteris H. Effectiveness of a modified Mother-Infant Transaction Program on outcomes for preterm infants from 3 to 24 months of age. Infant Behav Dev. 2009 Jan;32(1):17-26. doi: 10.1016/j.infbeh.2008.09.004. Epub 2008 Nov 20. PMID 19026450
- [Background] Bedrosian TA, Quayle C, Novaresi N, Gage FH. Early life experience drives structural variation of neural genomes in mice. Science. 2018 Mar 23;359(6382):1395-1399. doi: 10.1126/science.aah3378. PMID 29567711
- [Background] Ricci D, Romeo DM, Serrao F, Cesarini L, Gallini F, Cota F, Leone D, Zuppa AA, Romagnoli C, Cowan F, Mercuri E. Application of a neonatal assessment of visual function in a population of low risk full-term newborn. Early Hum Dev. 2008 Apr;84(4):277-80. doi: 10.1016/j.earlhumdev.2007.10.002. Epub 2007 Nov 8. PMID 17996405
- [Background] Guzzetta A, Baldini S, Bancale A, Baroncelli L, Ciucci F, Ghirri P, Putignano E, Sale A, Viegi A, Berardi N, Boldrini A, Cioni G, Maffei L. Massage accelerates brain development and the maturation of visual function. J Neurosci. 2009 May 6;29(18):6042-51. doi: 10.1523/JNEUROSCI.5548-08.2009. PMID 19420271